CLINICAL TRIAL: NCT01760655
Title: A Two Step Approach to Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for High Risk Hematologic Malignancies
Brief Title: Reduced-Intensity Conditioning Before Donor Stem Cell Transplant in With High-Risk Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12D.501; JT 2977 (Other: JeffTrial Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With Gene Mutations; Acute Myeloid Leukemia With Inv(3) (q21.3;q26.2); GATA2, MECOM; Acute Myeloid Leukemia With t(6;9) (p23;q34.1); DEK-NUP214; Aplastic Anemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Follicular Lymphoma; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloid Leukemia; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Polycythemia Vera; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Anemia, Aplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Leukemia, Myeloid; Lymphoma, Non-Hodgkin; Multiple Myeloma; Polycythemia Vera; Leukemia, Myeloid, Acute | interventions — fludarabine phosphate; Busulfan; methanesulfonic acid; Whole-Body Irradiation; Cyclophosphamide; Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (RIC and allogeneic PBSCT) (Experimental): REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV on days -15 to -12, busulfan IV on days -14 to -13, DLI on day -6, and cyclophosphamide IV on days -3 and -2. Patients also undergo TBI on day -10.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV on days -1 to 42 followed by taper and mycophenolate mofetil IV BID on days -1 to 28
  Interventions: Drug: Fludarabine phosphate; Drug: Busulfan; Radiation: Total-Body Irradiation; Biological: Therapeutic Allogeneic Lymphocytes; Drug: Cyclophosphamide; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; 75607-67-9; 9H-Purin-6-amine; 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; 2-fluoro-9-(5-O-phosphono-beta-D-arabinofuranosyl); Beneflur; Fludara; Fludarabine-5'-Monophosphate; SH T 586
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; 1,4-Bis(methanesulfonoxy)butane; 1,4-Bitanediol Dimethanesulfonate Esters; 1,4-Butanediol Dimethylsulfonate; 1,4-Di(methanesulfonyloxy)butane; 1,4-Di(methylsulfonyloxy)butane; 55-98-1; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid; tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; SCT_TBI; TOTAL BODY IRRADIATION; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Biological: Therapeutic Allogeneic Lymphocytes — Undergo DLI
  Other Names: Allogeneic Lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate; 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate; 2-[bis(b-chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane-2-oxide monohydrate; 2-[di(chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane 2-oxide monohydrate; 2H-1,3,2-Oxazaphosphorine; 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; 6055-19-2; bis(2-chloroethyl)phosphamide cyclic propanolamide ester monohydrate; Bis(2-chloroethyl)phosphoramide cyclic propanolamide ester monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; N,N-bis(2-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(2-chloroethyl)-N'-(3-hydroxypropyl)phosphorodiamidic acid intramolecular ester monohydrate; N,N-bis(2-chloroethyl)tetrahydro-2H-1,3,2-oxazaphosphorin-2-amine 2-oxide monohydrate; N,N-bis(b-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT; Stem Cell Transplantation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Drug: Tacrolimus — Given IV
  Other Names: 109581-93-3; FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Mycophenolate Mofetil — Given IV
  Other Names: 115007-34-6; 128794-94-5; Cellcept; MMF
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies reduced-intensity conditioning before donor stem cell transplant in treating patients with high-risk hematologic malignancies. Giving low-doses of chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) before the transplant may help increase this effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rate of disease-free survival (DFS) at 1 year post hematopoietic stem cell transplant (HSCT) in patients undergoing HSCT treated on this successor Thomas Jefferson University (TJU) 2 Step reduced intensity conditioning (RIC) haploidentical regimen and compare it with that of the initial 2 Step RIC regimen.

SECONDARY OBJECTIVES:

I. To assess the 100 day regimen-related mortality (RRM) in patients undergoing HSCT on this treatment protocol.

II. To determine the incidence and severity of graft-versus-host disease (GVHD) in patients undergoing treatment on this regimen.

III. To evaluate engraftment rates and lymphoid reconstitution in patients treated on this trial.

IV. To assess overall survival at 1 and 3 years past HSCT in patients treated on this trial.

OUTLINE:

REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) on days -15 to -12, busulfan IV on days -14 to -13, donor lymphocyte infusion (DLI) on day -6, and cyclophosphamide IV on days -3 and -2. Patients also undergo total-body irradiation (TBI) on day -10.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV on days -1 to 42 followed by taper and mycophenolate mofetil IV twice daily (BID) on days -1 to 28.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* By definition, patients with hematological malignancies or dyscrasias that require HSCT as part of cure-directed therapy are by definition high-risk and can be treated on this protocol; examples of high risk patients include but are not limited to:

  * Acute myeloid leukemia with high risk features as defined by:

    * Age greater than or equal to 60
    * Secondary acute myeloid leukemia (AML) (prior therapy or hematologic malignancy)
    * Normal cytogenetics but fms-related tyrosine kinase 3 (FLT3)/internal tandem duplication (ITD) positive
    * Any relapse or primary refractory disease
    * Greater than 3 cytogenetic abnormalities or any one of the following cytogenetic abnormalities: -5/del(5q), -7/del(7q), Abn(9q), (11q), (3q), (21q), (17p), t(6;9), t(6;11), t(11;19), +8, del(12p), inv(3), t(10;11), -17, 11q 23
    * Any single autosomal monosomy
  * Acute lymphoid leukemia in 1st or 2nd morphological remission; ALL with any morphological evidence of disease will not be eligible
  * Myelodysplasia (MDS) other than refractory anemia (RA), refractory anemia with rare sideroblasts (RARS), or isolated 5q- syndrome subtypes
  * Hodgkin's or Non-Hodgkin's lymphoma in 2nd or greater remission or with persistent disease
  * Myeloma with evidence of persistent disease after front-line therapy
  * Chronic myeloid leukemia (CML) resistant to signal transducer inhibitor (STI) therapy
  * Myelofibrosis and chronic myelomonocytic leukemia (CMML)
  * Essential thrombocytopenia or polycythemia vera with current or past evidence of evolution to acute leukemia
  * Patients with chronic lymphocytic leukemia (CLL), follicular non-Hodgkin lymphoma (NHL), or other lymphoid malignancies who have highly adverse cytogenetics (such as p53 deletion), are chemo-insensitive, are not responsive to highly effective novel treatments such as chimeric antigen receptor T-lymphocytes (CART) or Ibrutinib, or who have transformed disease
  * Any hematological malignancy not cited above which is thought to be high-risk with increased chance of post HSCT relapse
  * Any patient who has an aggressive disease that would normally be treated on a myeloablative study, but is prevented from doing so by factors in their past medical history; examples are patients with previous treatment with radiation therapy precluding TBI, or a past history of myeloablative therapy, precluding a 2nd myeloablative regimen
  * Patients with aplastic anemia may be treated on this protocol, with outcomes reported descriptively
* Patients must have a related donor who is at least a 2-4/8 antigen mismatch at the human leukocyte antigen (HLA)-A; B; C; DR loci; patients with only a 1 out of 8 mismatch in the GVH direction will be classified in the matched related category
* Left ventricular end diastolic function (LVEF) of >= 50%
* Diffusion lung capacity of oxygen (DLCO) >= 50% of predicted corrected for hemoglobin
* Serum bilirubin =< 1.8
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x upper limit of normal
* Creatinine clearance of >= 60 mL/min
* Patients < age 60 years must have a Karnofsky performance status (KPS) of >= 80% and a hematopoietic cell transplant comorbidity index (HCT-CI) score of 5 or less
* Patients aged 60 to 65 years must have a KPS of >= 80% and an HCT-CI score of 4 or less
* Patients aged 66 to 69 years must have a KPS of 90% and an HCT-CI score of 3 or less
* Patients aged 70 years or more must have a KPS of 90% and an HCT-CI score of 2 or less

  * (Patients with greater than the allowable HCT-CI points for age can be enrolled for trial with approval of the principal investigator [PI] and at least 1 co-investigator [Co-I] not on the primary care team of the patient) this is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than guideline HCT-CI points; an example is a patient with a solid tumor malignancy in their remote history (adds 3 points to HCT-CI total) where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities
* Patients must be willing to use contraception if they have childbearing potential
* Patient or patient's guardian is able to give informed consent

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive
* Active involvement of the central nervous system with malignancy; this can be documented as a normal neurological exam and/or a negative cerebrospinal fluid (CSF) analysis
* Pregnancy
* Patients with life expectancy of =< 6 months for reasons other than their underlying hematologic/oncologic disorder
* Patients who have received alemtuzumab or ATG within 8 weeks of the transplant admission
* Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12-24 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, RN, CRNP, DNP, Principal Investigator — Thomas Jefferson University; Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (RIC and allogeneic PBSCT): REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV on days -15 to -12, busulfan IV on days -14 to -13, DLI on day -6, and cyclophosphamide IV on days -3 and -2. Patients also undergo TBI on day -10.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV on days -1 to 42 followed by taper and mycophenolate mofetil IV BID on days -1 to 28
  Fludarabine phosphate: Given IV
  Busulfan: Given IV
  Total-Body Irradiation: Undergo TBI
  Therapeutic Allogeneic Lymphocytes: Undergo DLI
  Cyclophosphamide: Given IV
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSCT
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSCT
  Tacrolimus: Given IV
  Mycophenolate Mofetil: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Started | 62
Completed | 43
Not Completed | 19
Not completed — Death | 18
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: This hypothesis will be rejected if the 95% confidence interval for year DFS rate computed from the estimated Kaplan-Meier survival curves will be entirely above 0.35.
Time Frame: 1 year post hematopoietic stem cell transplant (HSCT)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 62
proportion of participants | .5 [.368 to .618]

2. Secondary Outcome: Overall Survival
Description: Will be analyzed and reported descriptively.
Time Frame: 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 62
proportion of participants | .567 [.432 to .681]

3. Secondary Outcome: Overall Survival
Description: Will be analyzed and reported descriptively.
Time Frame: 3 years post HSCT
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 62
proportion of participants | .479 [.347 to .599]

4. Secondary Outcome: Immune Reconstitution at Day +28
Description: CD4 and CD8 values at Day +28. Reported as mean (standard deviation).
Time Frame: Up to 1 year
Population: Participants surviving to Day +28 with evaluable data. This excludes the one subject who was a graft failure and anyone who died before 28 days.
Measure: Mean (Standard Deviation); unit: cells/mm³
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 56
cells/mm³
  CD3/4 at Day +28 | 66.9 (80.5)
  CD3/8 at Day +28 | 109.9 (137.4)

5. Secondary Outcome: Immune Reconstitution at Day +90
Description: CD4 and CD8 values at Day +90. Reported as mean (standard deviation).
Time Frame: Up to 1 year
Population: Participants surviving to Day +90 with evaluable data. This excludes the one subject who was a graft failure and anyone who died before 28 days.
Measure: Mean (Standard Deviation); unit: cells/mm³
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 44
cells/mm³
  CD3/4 at Day +90 | 173.7 (136.1)
  CD3/8 at Day +90 | 343.1 (395.4)

6. Secondary Outcome: Incidence and Degree of Graft Versus Host Disease
Description: The incidence and severity of graft-versus-host disease (GVHD) will be analyzed and reported descriptively. Clinical manifestations including skin rash, diarrhea, and liver function test abnormalities will be assessed. GVHD will be staged using established clinical grading systems: acute GVHD will be graded according to the modified Glucksberg criteria, and chronic GVHD will be graded using the NIH consensus criteria. These grading systems classify GVHD severity based on organ involvement and clinical symptoms. Higher stages or grades reflect more severe disease and are considered worse outcomes.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 59
Participants
  Grade 1 | 5
  Grade 2 | 15
  Grade 3 | 3
  Grade 4 | 3
  Missing/Cannot Assess | 2

7. Secondary Outcome: Engraftment Rates
Description: Will be analyzed and reported descriptively.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RIC and allogeneic PBSCT)
Number analyzed (Participants) | 60
Participants | 59

ADVERSE EVENTS:
Time Frame: All patients will be followed for adverse experiences (AEs) (serious and nonserious), regardless of relationships to study treatment, from the time of enrollment until d +100 after transplant
Arm/Group | Treatment (RIC and allogeneic PBSCT)
All-Cause Mortality (participants affected / at risk) | 27/62
Serious Adverse Events (participants affected / at risk) | 30/62
Other Adverse Events (participants affected / at risk) | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RIC and allogeneic PBSCT) (N=62)
Acute Kidney Injury - Grade 2 (Renal and urinary disorders) | 1 (1)
Acute Kidney Injury - Grade 4 (Renal and urinary disorders) | 2 (2)
Blood bilirubin increased - Grade 4 (Hepatobiliary disorders) | 1 (1)
Blood bilirubin increased - Grade 3 (Hepatobiliary disorders) | 1 (1)
cholelithiasis - grade 3 (Infections and infestations) | 1 (1)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fibrinogen - grade 4 (Blood and lymphatic system disorders) | 1 (1)
Heart failure - grade 3 (Cardiac disorders) | 2 (2)
Hypertension - Grade 4 (Cardiac disorders) | 2 (2)
Hypotension - Grade 4 (Cardiac disorders) | 1 (1)
Hypoxia - grade 3 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ileus - grade 3 (Gastrointestinal disorders) | 2 (2)
Infection - grade 3 (Infections and infestations) | 4 (4)
Infection - grade 4 (Infections and infestations) | 1 (1)
Infection - grade 1 (Infections and infestations) | 1 (1)
Infusion reaction - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Left ventricular systolic dysfunction - Grade 3 (Cardiac disorders) | 1 (1)
multi-organ failure - grade 4 (General disorders) | 2 (2)
Nausea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Opportunistic infection - grade 3 (Infections and infestations) | 2 (2)
Pain - Chest wall- grade 2 (Cardiac disorders) | 1 (1)
Pericardial effusion - Grade 4 (Cardiac disorders) | 1 (1)
Pulmonary edema - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
significant mucositis - grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — including tongue swelling and inability to clear secretions
Syncope - Grade 3 (Cardiac disorders) | 1 (1)
vasovagal episode - grade 3 (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RIC and allogeneic PBSCT) (N=62)
Abdominal Discomfort - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal Distention - Grade 1 (Gastrointestinal disorders) | 5 (5)
Acid Reflux - Grade 1 (Gastrointestinal disorders) | 1 (1)
Acute Kidney Injury - Grade 1 (Renal and urinary disorders) | 7 (7)
Acute Kidney Injury - Grade 2 (Renal and urinary disorders) | 1 (1)
Acute Kidney Injury - Grade 3 (Renal and urinary disorders) | 6 (6)
Acute Kidney Injury - Grade 4 (Renal and urinary disorders) | 3 (3)
Acute Pericatheter Thrombus - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Adenopathy - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation - Grade 2 (Cardiac disorders) | 4 (4)
Agitation - Grade 1 (Psychiatric disorders) | 1 (1)
Agitation - Grade 2 (Psychiatric disorders) | 3 (3)
Agitation - Grade 3 (Psychiatric disorders) | 1 (1)
Alanine Aminotransferase Levels Increased - Grade 3 (Hepatobiliary disorders) | 1 (1)
Alanine Aminotransferase Levels Increased - Grade 2 (Hepatobiliary disorders) | 1 (1)
Allergic Rhinitis - Grade 1 (Immune system disorders) | 2 (2)
Allergy To Amlodipine - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Allergy To Latex - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Alopecia - Grade 1 (Immune system disorders) | 12 (12)
Altered Mental State - Confusion - Grade 2 (Psychiatric disorders) | 1 (1)
Altered Taste - Grade 1 (General disorders) | 1 (1)
Anemia - Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Anger - Grade 1 (Psychiatric disorders) | 1 (1)
Anorexia - Grade 1 (Psychiatric disorders) | 3 (3)
Anorexia - Grade 2 (Psychiatric disorders) | 7 (7)
Anxiety - Grade 1 (Psychiatric disorders) | 12 (12)
Anxiety - Grade 2 (Psychiatric disorders) | 7 (7)
Aortic Aneurysm - Grade 1 (Cardiac disorders) | 1 (1)
Arthralgias - Grade 1 (Immune system disorders) | 6 (6)
Ascites - Grade 1 (Vascular disorders) | 1 (1)
Aspartate aminotransferase increased - Grade 2 (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased - Grade 3 (Hepatobiliary disorders) | 1 (1)
Asthma - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial fibrillation - Grade 1 (Cardiac disorders) | 1 (1)
Awakening To Urinate (Renal and urinary disorders) | 1 (1)
Bacteremia - Grade 2 (Infections and infestations) | 1 (1)
Bacteremia - Grade 3 (Infections and infestations) | 1 (1)
Benign Prostatic Hyperplasia - Grade 1 (Renal and urinary disorders) | 3 (3)
BK Cystitis - Grade 2 (Renal and urinary disorders) | 1 (1)
Bladder Spasm - Grade 1 (Renal and urinary disorders) | 1 (1)
Bleeding At Injection Sites - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Blister - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Blister - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Bloating - Grade 1 (Gastrointestinal disorders) | 2 (2)
Blood Bilirubin Increased - Grade 1 (Hepatobiliary disorders) | 1 (1)
Blood Bilirubin Increased - Grade 3 (Hepatobiliary disorders) | 4 (4)
Blurred Vision - Grade 1 (Eye disorders) | 2 (2)
Blurred Vision - Grade 2 (Eye disorders) | 1 (1)
Body Ache - Grade 1 (General disorders) | 1 (1)
Bradycardia - Grade 1 (Cardiac disorders) | 1 (1)
Bruising - Grade 1 (Vascular disorders) | 1 (1)
Painful Urination - Grade 1 (Renal and urinary disorders) | 1 (1)
Burning/Tearing of Eyes - Grade 1 (Eye disorders) | 1 (1)
Clostridioides Difficile Infection - Grade 1 (Infections and infestations) | 2 (2)
Cardiomyopathy - Grade 2 (Cardiac disorders) | 1 (1)
Colitis - Grade 1 (Infections and infestations) | 1 (1)
Cellulitis - Grade 1 (Infections and infestations) | 1 (1)
Change in Appetite/Weight Loss - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Change in Vision - Grade 1 (Eye disorders) | 1 (1)
Chest tightness - Grade 2 (General disorders) | 1 (1)
Chills - Grade 1 (General disorders) | 20 (20)
Chills - Grade 2 (General disorders) | 2 (2)
Choking - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic Constipation - Grade 1 (Gastrointestinal disorders) | 1 (1)
Chronic Hepatitis - Grade 1 (Renal and urinary disorders) | 1 (1)
Chronic Kidney Disease - Grade 1 (Renal and urinary disorders) | 1 (1)
Chronic Loose Stool - Grade 2 (Gastrointestinal disorders) | 1 (1)
COPD - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CMV Reactivation - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
CMV Reactivation - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cold Sweats - Grade 1 (General disorders) | 1 (1)
Colitis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Confusion - Grade 1 (Psychiatric disorders) | 4 (4)
Confusion - Grade 2 (Psychiatric disorders) | 1 (1)
Conjunctiva Hemorrhage - Grade 1 (Eye disorders) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 22 (22)
Constipation - Grade 2 (Gastrointestinal disorders) | 2 (2)
Coronary Artery Disease - Grade 1 (Vascular disorders) | 1 (1)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Cough - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine Increased - Grade 2 (Hepatobiliary disorders) | 1 (1)
Cytokine Release Syndrome - Grade 4 (Immune system disorders) | 1 (1)
Decreased Appetite - Grade 1 (Metabolism and nutrition disorders) | 17 (17)
Decreased Appetite - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Decreased Breath Sounds - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Concentration - Grade 1 (Psychiatric disorders) | 1 (1)
Decreased Ejection Fraction - Grade 1 (Cardiac disorders) | 1 (1)
Decreased Urine Output - Grade 1 (Renal and urinary disorders) | 5 (5)
Decreased Urine Output - Grade 2 (Renal and urinary disorders) | 1 (1)
Decreased White Blood Cell count - Grade 3 (Immune system disorders) | 1 (1)
Deep Vein Thrombosis - Grade 1 (Vascular disorders) | 2 (2)
Dehydration - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Dehydration - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Delirium - Grade 1 (Psychiatric disorders) | 1 (1)
Depressed Level of Consciousness - Grade 2 (Psychiatric disorders) | 1 (1)
Depression - Grade 1 (Psychiatric disorders) | 11 (11)
Depression - Grade 2 (Psychiatric disorders) | 4 (4)
Desquamation - Hands - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetes - Grade 1 (Metabolism and nutrition disorders) | 5 (5)
Diaphoresis - grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 33 (33)
Diarrhea - Grade 2 (Gastrointestinal disorders) | 10 (10)
Diarrhea - Grade 3 (Gastrointestinal disorders) | 9 (9)
Distension - Grade 1 (Gastrointestinal disorders) | 1 (1)
Distress - Grade 1 (Psychiatric disorders) | 1 (1)
Diverticulitis - Grade 2 (Gastrointestinal disorders) | 1 (1)
Dizziness - Grade 1 (General disorders) | 8 (8)
Dizziness - Grade 2 (General disorders) | 8 (8)
Dry eyes - Grade 1 (Eye disorders) | 2 (2)
Dry eyes - Grade 2 (Eye disorders) | 1 (1)
Dry Heaving - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dry Heaving -Grade 2 (Gastrointestinal disorders) | 1 (1)
Dry Mouth - Grade 1 (General disorders) | 9 (9)
Dry Mouth - Grade 2 (General disorders) | 2 (2)
Deep Vein Thrombosis - Grade 2 (Vascular disorders) | 3 (3)
Dysgeusia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dyslipidemia - Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Dyslipidemia - Grade 2 (Blood and lymphatic system disorders) | 1 (1)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dysphagia - Grade 1 (Musculoskeletal and connective tissue disorders) | 4 (4)
Dysphagia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea on Exertion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysuria - Grade 1 (Renal and urinary disorders) | 9 (9)
Dysuria - Grade 3 (Renal and urinary disorders) | 1 (1)
Ecchtmosis - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
E-coli Infection - Grade 1 (Infections and infestations) | 1 (1)
Eczema - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Edema - Grade 1 (Vascular disorders) | 21 (21)
Edema - Grade 2 (Vascular disorders) | 9 (9)
Skin Tears - Elbow - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Electrolyte Imbalance - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Electrolyte Imbalance - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Elevated Bilirubin - Grade 2 (Hepatobiliary disorders) | 1 (1)
Elevated Liver Function Tests - Grade 1 (Hepatobiliary disorders) | 3 (3)
Encephalopathy - Grade 1 (Nervous system disorders) | 1 (1)
Encephalopathy - Grade 4 (Nervous system disorders) | 1 (1)
Epistaxis - Grade 1 (Skin and subcutaneous tissue disorders) | 6 (6)
Erectile Dysfunction - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Extremity Weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 5 (5)
Eye Problems - Grade 1 (Eye disorders) | 1 (1)
Facial Puffiness - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Flushing - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
Failure to Thrive - Grade 1 (General disorders) | 1 (1)
Fall - Grade 1 (Injury, poisoning and procedural complications) | 5 (5)
Fall - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Fatigue - Grade 1 (General disorders) | 26 (26)
Fatigue - Grade 2 (General disorders) | 3 (3)
Fatigue - Grade 3 (General disorders) | 6 (6)
Fever - Grade 1 (Immune system disorders) | 43 (43)
Fever - Grade 2 (Immune system disorders) | 8 (8)
Fever - Grade 3 (Immune system disorders) | 7 (7)
Flatulence - Grade 1 (Gastrointestinal disorders) | 4 (4)
Floaters - grade 1 (Eye disorders) | 1 (1)
Folliculitis - grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Gait Disturbance - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Body Aches - Generalized (General disorders) | 1 (1)
GERD - Grade 1 (Gastrointestinal disorders) | 1 (1)
GERD - Grade 2 (Gastrointestinal disorders) | 2 (2)
GERO - Grade 1 (Gastrointestinal disorders) | 5 (5)
Gouty Changes in Digits (Musculoskeletal and connective tissue disorders) | 2 (2)
Hallucinations - Grade 1 (Psychiatric disorders) | 6 (6)
Hallucinations - Grade 2 (Psychiatric disorders) | 1 (1)
Headache - Grade 1 (General disorders) | 17 (17)
Headache - Grade 2 (General disorders) | 5 (5)
Headache - Grade 3 (General disorders) | 1 (1)
Hearing Loss - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Heart Murmur - Grade 1 (Cardiac disorders) | 1 (1)
Heartburn - Grade 1 (Gastrointestinal disorders) | 1 (1)
Hematuria - Grade 1 (Renal and urinary disorders) | 10 (10)
Hematuria - Grade 2 (Renal and urinary disorders) | 5 (5)
Hemmorhoidal Bleeding - Grade 1 (Vascular disorders) | 1 (1)
Hemolytic Uremic Syndrome - Grade 5 (Blood and lymphatic system disorders) | 1 (1)
Hemorrhoids - Grade 1 (Vascular disorders) | 4 (4)
Hemorrhoids - Grade 2 (Vascular disorders) | 1 (1)
HHV-6 Viremia - Grade 1 (Infections and infestations) | 2 (2)
Hives - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hoarseness - Grade 1 (General disorders) | 2 (2)
Hyperbilirubin - Grade 1 (Hepatobiliary disorders) | 3 (3)
Hyperbilirubinemia - Grade 2 (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinemia - Grade 4 (Hepatobiliary disorders) | 1 (1)
Hypercalcemia - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Hyperlipidemia - Grade 1 (Blood and lymphatic system disorders) | 5 (5)
Hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension - Grade 1 (Vascular disorders) | 21 (21)
Hypertension - Grade 2 (Vascular disorders) | 9 (9)
Hypertension - Grade 3 (Vascular disorders) | 2 (2)
Hypervolemia - Grade 2 (Vascular disorders) | 3 (3)
Hypervolemia - Grade 2 (Blood and lymphatic system disorders) | 7 (7)
Hyperkalemia - Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Hypomagnesemia - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Hypotension - Grade 1 (General disorders) | 17 (17)
Hypotension - Grade 2 (Vascular disorders) | 8 (8)
Hypotension - Grade 4 (Vascular disorders) | 2 (2)
Hypothyroidism - Grade 1 (Endocrine disorders) | 1 (1)
Hypoxia - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Hypoxia - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus - Grade 3 (Gastrointestinal disorders) | 1 (1)
Impaired Skin Integrity - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Increase of Right Atrial Pressure - Grade 1 (Cardiac disorders) | 1 (1)
Increased Creatinine - Grade 1 (Hepatobiliary disorders) | 2 (2)
Increased Creatinine - Grade 3 (Hepatobiliary disorders) | 1 (1)
Indigestion - Grade 1 (Gastrointestinal disorders) | 2 (2)
Infection (Other) - Grade 3 (Infections and infestations) | 4 (4)
Infusion Reaction - Grade 1 (Injury, poisoning and procedural complications) | 4 (4)
Infusion Reaction - Grade 2 (Injury, poisoning and procedural complications) | 7 (7)
Insomnia - Grade 1 (Psychiatric disorders) | 21 (21)
Insomnia - Grade 2 (Psychiatric disorders) | 4 (4)
Jaw Swelling - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Laryngitis - Grade 1 (General disorders) | 1 (1)
Left Ventricular Dysfunction - grade 3G (Cardiac disorders) | 1 (1)
Leg Cramps - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Lethargy - Grade 1 (General disorders) | 7 (7)
Lethargy - Grade 2 (General disorders) | 1 (1)
Low fibrinogen - Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Parotitis - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Orthostatic Hypotension - Grade 1 (Cardiac disorders) | 1 (1)
PACs - Grade 1 (Cardiac disorders) | 1 (1)
Palpitations - Grade 1 (Cardiac disorders) | 2 (2)
Palpitations - Grade 2 (Cardiac disorders) | 1 (1)
Pericardial Effusion - Grade 1 (Cardiac disorders) | 1 (1)
Pericardial Effusion - Grade 3 (Cardiac disorders) | 1 (1)
Pericardial Effusion - Grade 4 (Cardiac disorders) | 1 (1)
Sinus Bradycardia - Grade 1 (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia - Grade 1 (Cardiac disorders) | 1 (1)
Tachycardia - Grade 3 (Cardiac disorders) | 1 (1)
Ventricular Tachycardia - Grade 2 (Cardiac disorders) | 1 (1)
Pericardial Effusion - Grade 2 (Cardiac disorders) | 2 (2)
Tachycardia - Grade 2 (Cardiac disorders) | 3 (3)
Premature Ventricular Contractions - Grade 1 (Cardiac disorders) | 4 (4)
Tachycardia - Grade 1 (Cardiac disorders) | 21 (21)
Tinnitus - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Visual Disturbance - Grade 1 (Eye disorders) | 2 (2)
Puffy Eyes -Grade 1 (Eye disorders) | 1 (1)
Retinal Detachment - Grade 3 (Eye disorders) | 1 (1)
Right Eye Irritation/Tearing - Grade 2 (Eye disorders) | 1 (1)
Scleral Edema - Grade 1 (Eye disorders) | 1 (1)
Scleral Injection - Grade 1 (Eye disorders) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 20 (20)
Red Macule on Uvula - Grade 1 (Gastrointestinal disorders) | 1 (1)
Soreness - Grade 1 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 1 (Gastrointestinal disorders) | 20 (20)
Nausea - Grade 2 (Gastrointestinal disorders) | 10 (10)
Vomiting - Grade 2 (Gastrointestinal disorders) | 6 (6)
Malnutrition - Grade 3 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 3 (Gastrointestinal disorders) | 1 (1)
Pain - Grade 1 (General disorders) | 1 (1)
Pain (Esophageal) - Grade 1 (General disorders) | 1 (1)
Pain (Flank) - Grade 1 (General disorders) | 1 (1)
Pain (Jaw) - Grade 1 (General disorders) | 1 (1)
Pain (Left Extremities) - Grade 1 (General disorders) | 1 (1)
Pain (Left Flank) - Grade 1 (General disorders) | 1 (1)
Pain (Leg) - Grade 1 (General disorders) | 1 (1)
Pain (Lower Quadrant) - Grade 1 (General disorders) | 1 (1)
Pain (Mouth) - Grade 1 (General disorders) | 1 (1)
Pain (Perianal) - Grade 1 (General disorders) | 1 (1)
Pain (Rib) - Grade 1 (General disorders) | 1 (1)
Pain (Toe) - Grade 1 (General disorders) | 1 (1)
Pain (Tooth) - Grade 1 (General disorders) | 1 (1)
Painful Swallowing - Grade 1 (General disorders) | 1 (1)
Pleuritic Pain - Grade 1 (General disorders) | 1 (1)
Problems with Balance/ Dizziness - Grade 1 (General disorders) | 1 (1)
Pain (Arm) - Grade 1 (General disorders) | 2 (2)
Pain (Foot) - Grade 1 (General disorders) | 2 (2)
Pain (Gastrointenstinal) - Grade 1 (General disorders) | 2 (2)
Pain (Rectal) - Grade 1 (General disorders) | 2 (2)
Pain (Scrotal) - Grade 1 (General disorders) | 2 (2)
Myalgias - Grade 1 (General disorders) | 3 (3)
Rigors - Grade 1 (General disorders) | 3 (3)
Sore Throat - Grade 1 (General disorders) | 3 (3)
Pain (Shoulder) - Grade 1 (General disorders) | 6 (6)
Pain (Chest) - Grade 1 (General disorders) | 6 (6)
Weakness - Grade 1 (General disorders) | 7 (7)
Lightheadedness - Grade 1 (General disorders) | 9 (9)
Pain (Abdominal) - Grade 1 (General disorders) | 14 (14)
Pain (Back) - Grade 1 (General disorders) | 12 (12)
Malaise - Grade 2 (General disorders) | 1 (1)
Pain (General) - Grade 2 (General disorders) | 1 (1)
Pain (Hemorrhoids) - Grade 2 (General disorders) | 1 (1)
Pain (Jaw) - Grade 2 (General disorders) | 1 (1)
Pain (Joint/Muscle) - Grade 2 (General disorders) | 1 (1)
Pain (Leg) - Grade 2 (General disorders) | 1 (1)
Pain (Perianal) - Grade 2 (General disorders) | 1 (1)
Pain (Sciatica) - Grade 2 (General disorders) | 1 (1)
Pain (Shoulder) - Grade 2 (General disorders) | 1 (1)
Sore Throat - Grade 2 (General disorders) | 1 (1)
Weakness - Grade 2 (General disorders) | 1 (1)
Pain (Abdominal) - Grade 2 (General disorders) | 3 (3)
Pain (Back) - Grade 2 (General disorders) | 2 (2)
Pain (Buttock) - Grade 2 (General disorders) | 2 (2)
Pain (Chest) - Grade 2 (General disorders) | 2 (2)
Weakness - Grade 3 (General disorders) | 1 (1)
Nasal Congestion - Grade 1 (Immune system disorders) | 3 (3)
Osteoarthritis - Grade 1 (Immune system disorders) | 1 (1)
Post Nasal Drip - Grade 1 (Immune system disorders) | 1 (1)
Rheumatoid Arthritis - Grade 1 (Immune system disorders) | 1 (1)
Rhinorrhea - Grade 1 (Immune system disorders) | 2 (2)
Sinusitis - Grade 1 (Immune system disorders) | 1 (1)
Sneezing - Grade 1 (Immune system disorders) | 1 (1)
Sinusitis - Grade 2 (Immune system disorders) | 1 (1)
Sinusitis - Grade 3 (Immune system disorders) | 1 (1)
Oral Thrush - Grade 1 (Infections and infestations) | 1 (1)
Rhinovirus -Grade 1 (Infections and infestations) | 1 (1)
Pneumonia - Grade 2 (Infections and infestations) | 1 (1)
Thrush - Grade 2 (Infections and infestations) | 3 (3)
Vaginitis - Grade 2 (Infections and infestations) | 1 (1)
Periorbital Infection - Grade 3 (Infections and infestations) | 1 (1)
Sepsis - Grade 4 (Infections and infestations) | 1 (1)
Sepsis - Grade 5 (Infections and infestations) | 1 (1)
Pericatheter Thrombus - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Skin Wound - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Metabolic Syndrome - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Obesity - Grade 1 (Metabolism and nutrition disorders) | 6 (6)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Weight Gain - Grade 1 (Metabolism and nutrition disorders) | 3 (3)
Weight Gain - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Weight Loss - Grade 1 (Metabolism and nutrition disorders) | 6 (6)
Thrombus - Grade 1 (Vascular disorders) | 1 (1)
Thrombotic Microangiopathy - Grade 2 (Vascular disorders) | 1 (1)
Thromboembolic Event - Grade 2 (Vascular disorders) | 3 (3)
Syncope - Grade 3 (Vascular disorders) | 4 (4)
Lower Extremity Weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Cramping - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy - Grade 1 (Musculoskeletal and connective tissue disorders) | 9 (9)
Paresthesia - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Singultus - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Tremor - Grade 1 (Musculoskeletal and connective tissue disorders) | 5 (5)
Neuropathy - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Singultus - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis - Grade 1 (Skin and subcutaneous tissue disorders) | 7 (7)
Night Sweats - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Peeling lips - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Penile Swelling - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral Edema - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash-Maculo-Papular - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Right Buttock Wound - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Right Heel Skin Tear - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp Sensitivity - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Tear on Scrotum - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Tenosynovitis of Ankle - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Ulcer on Right Ankle - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal Irritation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Photophobia - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Scrotal Edema - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 15 (15)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 31 (31)
Mucositis - Grade 2 (Skin and subcutaneous tissue disorders) | 4 (4)
Peripheral Edema - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 9 (9)
Scrotal Edema - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Scrotal Irritation - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal Hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis - Grade 3 (Skin and subcutaneous tissue disorders) | 20 (20)
Rash - Grade 3 (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal Hemorrhage - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Obstructive Sleep Apnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchi - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep Apnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Tachypnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Shortness of Breath - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pleural Effusion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary Congestion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachypnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, Thorasic and Mediastinal Disorders (Other) - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnea - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nocturia - Grade 1 (Renal and urinary disorders) | 5 (5)
Polyuria - Grade 1 (Renal and urinary disorders) | 2 (2)
Urgency of Urine - Grade 2 (Renal and urinary disorders) | 2 (2)
Urinary Frequency - Grade 1 (Renal and urinary disorders) | 10 (10)
Urinary Incontinence - Grade 1 (Renal and urinary disorders) | 5 (5)
Urinary Retention - Grade 1 (Renal and urinary disorders) | 2 (2)
Urinary Tract Infection - Grade 1 (Renal and urinary disorders) | 1 (1)
Obstructive Sleep Apnea - Grade 2 (Renal and urinary disorders) | 1 (1)
Proteinuria - Grade 2 (Renal and urinary disorders) | 2 (2)
Renal Insufficiency - Grade 2 (Renal and urinary disorders) | 1 (1)
Urinary Pain - Grade 2 (Renal and urinary disorders) | 1 (1)
Urine Output Decreased - Grade 3 (Renal and urinary disorders) | 1 (1)
Suicidal Ideation - Grade 1 (Psychiatric disorders) | 1 (1)
Speech or Memory Change - Grade 1 (Psychiatric disorders) | 1 (1)
Racing Thoughts - Grade 1 (Psychiatric disorders) | 1 (1)
Panic Attack - Grade 2 (Psychiatric disorders) | 1 (1)
Mental Status Change - Grade 2 (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT01760655/Prot_SAP_000.pdf